CLINICAL TRIAL: NCT02709811
Title: Safety and Feasibility of Electrochemotherapy in the Treatment of Unresectable Liver Metastases From Colorectal Adenocarninoma
Brief Title: Safety and Feasibility of Electrochemotherapy in Unresectable Colorectal Adenocarninoma Liver Metastases
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment at study center below rate compatible with study completion.
Sponsor: IGEA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PECTL1
Record Dates: First submitted 2014-11-24; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Adenocarcinoma
MeSH Terms: interventions — Electrochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- electrochemotherapy (Experimental)
  Interventions: Drug: Electrochemotherapy

INTERVENTIONS:
Drug: Electrochemotherapy

SUMMARY:
Electrochemotherapy (ECT) is a non-thermal tumour ablation modality. It consists of the local potentiation, by means of local reversible electroporation of tumour tissues, of the antitumor activity of non-permeant or poorly permeant anticancer drugs already possessing intrinsic cytotoxicity. ECT has proved to be effective in the treatment of various cutaneous tumour nodules of any origin. Mostly ECT is offered to patients in case of multiple cutaneous metastases, when they cannot be excised, due to their number or localization. This study investigate the application of ECT in the treatment of liver metastases from colorectal adenocarcinoma, for which other thermal cytoreductive methods would be risky compared to the supposed expected clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years of age
* Histological confirmed colorectal adenocarcinoma
* Histological or clinically confirmed metastatic colorectal adenocarcinoma lesions (liver lesions only are considered as metastatic disease) and not resecable.
* A single liver lesion may not exceed 3 cm
* Liver lesions must not have a depth greater than 2 cm from hepatic surface (Glisson Capsule) (measured clinically if possible otherwise on the basis of CT/ultrasound examination)
* A life expectancy of at least 6 months.
* Patients with a ECOG performance status < 2
* Signed Informed Consent
* Patient must be mentally capable of understanding the information given.
* Patient must give informed consent.

Exclusion Criteria:

* Age less than 18 years.
* Patient pregnant or lactating (no contraceptive method is contraindicated, a pregnancy test will be administered to all women of childbearing age)
* Life-threatening infection and/or heart failure and/or liver failure and/or other severe systemic pathologies that preclude laparotomy
* Strumental analysis confirmed ascites.
* Impaired kidney function.
* Significant reduction in respiratory function.
* Allergic reaction to bleomycin.
* Coagulation disturbances
* Patients with exclusion criteria for diagnostic MRI 3Tesla (with pace-makers and all those metal devices that are not compatible with 3T).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility evaluation of Electrochemotherapy treatment of liver metastasesSafety and feasibility evaluation of Electrochemotherapy treatment of liver metastases as meaured by unexpected intraoperative adverse events | 24 hours from Electrochemotherapy treatment
  Safety and feasibility evaluation of Electrochemotherapy treatment of liver metastases as meaured by unexpected intraoperative adverse events and related postoperative complications.

SECONDARY OUTCOMES:
Overall survival | 6 months from Electrochemotherapy treatment
Disease free survival | 6 months from Electrochemotherapy treatment
Quality of Life (Karnofsky performance status) | 30 days and 6 months from ECT treatment
Objective response evaluation of treated liver metastases following RECIST criteria | 30 days and 6 months from Electrochemotherapy treatment
Toxicity of Electrochemotherapy treatment of liver metastases as meaured by unexpected postoperative complications related to treatment | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Franco Filipponi, MD, Principal Investigator — University of Pisa Medical School Hospital, Pisa, Italy